CLINICAL TRIAL: NCT06451549
Title: Real-world Evaluation of a Recommender System for Mental Health Self-management
Brief Title: Clinical Investigation of Syndi
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been withdrawn due to significant changes in its scope, which no longer align with the original protocol.
Sponsor: Newcastle University (Other)
Collaborators: Cornwall Partnership NHS Foundation Trust (Network); University of Plymouth (Other)
Responsible Party: Principal Investigator, Edward Meinert, Professor of Digital Health and Clinical Artificial Intelligence, Newcastle University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU-015775
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Mental Health Issue; Depression; Anxiety
Keywords: Digital Health; Recommender System; Mental Health; Telemedicine
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: All participants will be given access to Syndi immediately
Masking Description: As this is a single arm study, all participants will receive the intervention and no masking is required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Syndi recommender system for mental health apps (Experimental): Syndi is a recommender system for mental health apps, delivered via a website. It guides users through a clinically-validated self-assessment and uses a machine learning system to provide personalised recommendations of independently-rated mental health tools.
  Interventions: Device: Syndi recommender system for mental health apps

INTERVENTIONS:
Device: Syndi recommender system for mental health apps — Syndi is a mental health app recommendation system. It provides personalised suggestions of apps to help users self-manage their mental health based on a clinical assessment.

SUMMARY:
Mental health concerns are a growing global concern, but support can still be difficult to access. Digital health technologies can help people access support, but with over 10,000 mental health apps available, it can be difficult to choose one that is safe, effective, and personalised. Syndi is a digital health platform that uses a machine learning system to provide personalised recommendations of mental health apps. This study aims to examine the impact of Syndi and its recommendations on the mental health and well-being of people with mental health concerns.

The investigators will use the standard National Health Service (NHS) Talking Therapies measures of anxiety and depression, as well as additional measures of wellbeing and functional impairment to look at the impact of Syndi on patients' mental well-being. The investigators will also look at user experience with Syndi using a survey. Users' engagement with Syndi and its recommended apps will be assessed using a short survey and some participants will be randomly selected for an interview so the investigators can get a better understanding of what people liked and disliked about using the platform and why.

The investigators expect that the project will show that using Syndi helps improve mental well-being in people with mental health concerns. If the study shows this positive impact, this will provide evidence to support the use of Syndi to improve the accessibility of mental health support in clinical pathways. The investigators will publish the results of the study in academic journals as well as in more accessible platforms.

ELIGIBILITY:
Inclusion Criteria:

* Based in the UK
* Referred or self-referred to proceed through the standard NHS Talking Therapies care pathway OR people with mental health concerns looking for app recommendations online;
* Willing and able to provide informed consent;
* Aged 18 years or older;
* Able to speak English;
* Have access to the internet and own a smartphone.

Exclusion Criteria:

* Patients with a PHQ-9 score >=20
* Patients with suicidal ideation measured as an answer of 'YES' to any question in the Columbia Suicide Severity Rating Scale (C-SSRS);
* Incapable of self-consent;
* In a dependent/unequal relationship with the research or care teams or any PPI representatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Depression Severity | 2 weeks and 3 months post-baseline
  Score on the Patient Health Questionnaire-9 (PHQ-9), total scores range from 0 to 27 (higher scores indicate more severe depression)

SECONDARY OUTCOMES:
Anxiety Severity | 2 weeks and 3 months post-baseline
  Score on the Generalised Anxiety Disorder-7 (GAD-7), total scores range from 0 to 21 (higher scores indicate more severe anxiety)
Mental Wellbeing | 2 weeks and 3 months post-baseline
  Score on the Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS), total scores range from 7 to 35 (higher scores indicate better wellbeing)
Functional Impairment | 2 weeks and 3 months post-baseline
  Score on the Work and Social Adjustment Scale (WSAS), total scores range from 0 to 40 (higher scores indicate higher functional impairment)
Engagement with recommended apps | 2 weeks post-baseline
  Self-report questionnaire about engagement with recommended apps (subjective, with questions about which apps were downloaded, how long they used it for, and how useful they found the app)
User experience with the Syndi recommender system | Immediately after app recommendations and at 2 weeks post-baseline
  Score on a user experience questionnaire. Items were assessed individually on a scale from 1-5, with higher scores indicating better experience (negative items were reverse coded)
User perceptions of the system | Semi-structured interview call, 2 months after start of the trial
  Qualitative feedback from semi-structured interviews about Syndi
User perceptions of the recommended apps | Semi-structured interview call, 2 months after start of the trial
  Qualitative feedback from semi-structured interviews about the apps recommended by Syndi

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Shankar, FRPsych, Principal Investigator — University of Plymouth
Locations (4):
- United Kingdom (4):
  - Pennine Care NHS Foundation Trust, Ashton-under-Lyne, Lancashire
  - Newcastle University, Newcastle upon Tyne, Tyne and Wear
  - Cornwall Partnership NHS Foundation Trust, Bodmin
  - Devon Partnership NHS Trust, Exeter

IPD SHARING:
Plan to Share IPD: No
Only the Academic CIs and their research staff will have access to research data.